CLINICAL TRIAL: NCT01873586
Title: Efficacy and Safety of OsteoStrux™ Collagen Ceramic Scaffold in Instrumented Lumbar Spine Fusion
Brief Title: OsteoStrux™ Collagen Ceramic Scaffold in Instrumented Lumbar Spine Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SeaSpine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OSX-US-2012-1
Record Dates: First submitted 2013-05-24; First posted 2013-06-10 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Degenerative Changes; Stenosis; Spondylosis
MeSH Terms: conditions — Constriction, Pathologic; Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OsteoStrux Collagen Ceramic Scaffold (Experimental): OsteoStrux Collagen Ceramic Scaffold (posterolateral gutter at the symptomatic side)
  Interventions: Procedure: Posterolateral Fusion
- Local autograft (Active Comparator): Local autograft (posterolateral gutter at the contralateral side)
  Interventions: Procedure: Posterolateral Fusion

INTERVENTIONS:
Procedure: Posterolateral Fusion

SUMMARY:
The objective of this study is to prospectively evaluate the performance of Integra's OsteoStrux Collagen Ceramic Scaffold combined with bone marrow aspirate as an adjunct for instrumented posterolateral spine fusion, as compared to local autograft.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 (eighteen) years of age or older at the time of surgery.
2. Require spinal fusion using TLIF, PLF or PLIF, with or without the use of an interbody spacer, at 1 to 3 levels between L3-S1.
3. Are willing and able to return for the scheduled follow-up visits, follow post-operative instructions and undergo the required radiographic exams (A/P, Lateral Neutral and Lateral Flexion/Extension X-rays) for up to 4 time points between 3 weeks and 12 months post-surgery (3 months ± 2 weeks, 6±1 months, 12±2 months and if required 24±3 months post-surgery), including one CT-scan at 12±2 months.
4. Are unresponsive to conservative care over a period of at least 6 months or have signs and/or symptoms that mandate urgent surgical intervention.
5. Are willing and able to sign study specific informed consent.

Exclusion Criteria:

1. Are long term users of medications (i.e. steroids greater than 8 days) that are known to inhibit fusion or bone metabolism at any time within 6 months prior to surgery. Exceptions are inhaled steroids for asthma treatment (i.e. patients on inhaled steroids are allowed), or epidural steroid injections.
2. Are taking immunosuppressive agents (Cancer chemotherapy, treatment with Disease Modifying Anti-rheumatic drugs (DMARDs) or any similar immunomodulating drugs) or are treated with Growth Factors or Insulin at any time within 6 months prior to surgery.
3. Are being treated with radiotherapy.
4. Are having medical conditions, known to impact bone metabolism, such as Paget's disease, or has established osteoporosis (i.e. has had one or more fragility fractures).
5. Are pregnant, lactating or women wishing to become pregnant.
6. Are a prisoner.
7. BMI ≥ 40
8. Are smokers and/or nicotine/tobacco users
9. Are currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the study endpoints.
10. Had prior spine surgery at the index level except posterior decompressive surgery where the posterior elements are preserved e.g. facet saving techniques such as discectomy, laminotomy, and intradiscal procedures.
11. Use of routine prophylactic NSAIDS for 3 months post-operatively, but low dose concomitant pain medications e.g. aspirin should be continued and recorded on the Concomitant Pain Medications case report form (CRF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Sherban, DO, Principal Investigator — Sherban Orthopaedic and Spine Surgery, PLLC
Locations (1):
- Sherban Orthopaedic and Spine Surgery, PLLC, Kenmore, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Posterolateral fusion study in which each patient undergoes posterolateral fusion. During the posterolateral fusion, each spinal level is treated with two grafts, the symptomatic posterolateral gutter is treated with study arm (OsteoStrux) and the contralateral posterolateral gutter is treated with the control arm (local autograft).
Units Other Than Participants: Spinal Levels
Groups:
- All Patients: Posterolateral fusion study in which each patient undergoes posterolateral fusion. During the posterolateral fusion, each spinal level is treated with two grafts, the symptomatic posterolateral gutter is treated with study arm (OsteoStrux) and the contralateral posterolateral gutter is treated with the control arm (local autograft).
Period: Overall Study
Arm/Group | All Patients
Started | 29; 54 Spinal Levels
Completed | 26; 47 Spinal Levels
Not Completed | 3; 7 Spinal Levels
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Posterolateral fusion study in which each patient undergoes posterolateral fusion. During the posterolateral fusion, each spinal level is treated with two grafts, the symptomatic posterolateral gutter is treated with study arm (OsteoStrux) and the contralateral posterolateral gutter is treated with the control arm (local autograft).
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: years] | 57 [31 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Posterolateral Gutters That Have Evidence of Arthrodesis (Fusion) at 3, 6, 12, and 24 Months, as Measured by X-rays.
Description: Posterolateral fusion study in which each patient undergoes posterolateral fusion. During the posterolateral fusion, each spinal level is treated with two grafts, the symptomatic posterolateral gutter is treated with study arm (OsteoStrux) and the contralateral posterolateral gutter is treated with the control arm (local autograft).
Time Frame: up to 24 months
Population: Posterolateral fusion study in which each patient undergoes posterolateral fusion. During the posterolateral fusion, each spinal level is treated with two grafts, the symptomatic posterolateral gutter is treated with study arm (OsteoStrux) and the contralateral posterolateral gutter is treated with the control arm (local autograft).
Measure: Count of Units; unit: Posterolateral Gutters
Units Other Than Participants: Posterolateral Gutters
Arm/Group | All Patients
Number analyzed (Participants) | 29
Number analyzed (Posterolateral Gutters) | 54
Posterolateral Gutters
  3 Month: OsteoStux (symptomatic): number analyzed (Participants) | 24
  3 Month: OsteoStux (symptomatic): number analyzed (Posterolateral Gutters) | 42
  3 Month: OsteoStux (symptomatic) | 39
  3 Month: Local Autograft (contralateral): number analyzed (Participants) | 25
  3 Month: Local Autograft (contralateral): number analyzed (Posterolateral Gutters) | 42
  3 Month: Local Autograft (contralateral) | 34
  6 Month: OsteoStux (symptomatic): number analyzed (Participants) | 25
  6 Month: OsteoStux (symptomatic): number analyzed (Posterolateral Gutters) | 46
  6 Month: OsteoStux (symptomatic) | 42
  6 Month : Local Autograft (contralateral): number analyzed (Participants) | 25
  6 Month : Local Autograft (contralateral): number analyzed (Posterolateral Gutters) | 46
  6 Month : Local Autograft (contralateral) | 36
  12 Month: OsteoStux (symptomatic): number analyzed (Participants) | 26
  12 Month: OsteoStux (symptomatic): number analyzed (Posterolateral Gutters) | 47
  12 Month: OsteoStux (symptomatic) | 44
  12 Month: Local Autograft (contralateral): number analyzed (Participants) | 26
  12 Month: Local Autograft (contralateral): number analyzed (Posterolateral Gutters) | 47
  12 Month: Local Autograft (contralateral) | 32
  24 Month: OsteoStux (symptomatic): number analyzed (Participants) | 26
  24 Month: OsteoStux (symptomatic): number analyzed (Posterolateral Gutters) | 47
  24 Month: OsteoStux (symptomatic) | 43
  24 Month: Local Autograft (contralateral): number analyzed (Participants) | 26
  24 Month: Local Autograft (contralateral): number analyzed (Posterolateral Gutters) | 47
  24 Month: Local Autograft (contralateral) | 34

2. Secondary Outcome: Number of Posterolateral Gutters Showing Evidence of Arthrodesis (Fusion) as Measured by CT
Description: Each posterolateral gutter was assessed for extent of fusion using computed tomography (CT) scan.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Units; unit: Posterolateral gutters
Units Other Than Participants: Posterolateral gutters
Arm/Group | All Patients
Number analyzed (Participants) | 25
Number analyzed (Posterolateral gutters) | 45
Posterolateral gutters
  12 Months: OsteoStrux (symptomatic) | 39
  12 Months: Local Autograft (contralateral) | 32

3. Secondary Outcome: Interbody Fusion as Determined by X-ray at 3, 6, 12 and 24 Months
Description: NA (Not Applicable): This post-market study was primarily a posterolateral fusion study. Interbody fusion was a secondary endpoint. As interbody fusion was completed per standard of care, transforaminal lumbar interbody fusion (TLIF), posterolateral fusion (PLF), or posterior lumbar interbody fusion (PLIF) with or without the use of an interbody spacer and any graft material could be used per the Investigator discretion. As interbody fusion was indistinguishable per arms, data were not collected due to a limitation in the method of analysis per protocol. Therefore data was not analyzed and outcome is NA.
Time Frame: upto 24 months
Population: NA (Not Applicable): As interbody fusion was not a primary endpoint and was indistinguishable per control and study arms, interbody fusion results were not analyzed.
Arm/Group | All Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Interbody Fusion as Determined by CT Post-surgery at Available Time-points
Description: NA (Not Applicable): This post-market study was primarily a posterolateral fusion study. Interbody fusion was a secondary endpoint. As interbody fusion was completed per standard of care, transforaminal lumbar interbody fusion (TLIF), posterolateral fusion (PLF), or posterior lumbar interbody fusion (PLIF) with or without the use of an interbody spacer and any graft material could be used per the Investigator discretion. As interbody fusion was not a primary endpoint and was indistinguishable per control and study arms, interbody fusion results were not analyzed.
Time Frame: 12 months
Population: as for outcome 3
Arm/Group | All Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: EQ-5D Health State Visual Analog Scale (VAS) Questionnaire at All Available Time-points
Description: EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS. The EQ-5D-5l has a descriptive system and the EQ visual analogue scale (EQ VAS).The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels which results in a 1-5 level selected for that dimension. The level when added together describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. Score is 0-100 and a lower score represents a better score.
Time Frame: upto 24 months
Population: Posterolateral fusion study in which one level is treated with both the study and control arm. One side is OsteoStrux combined with bone marrow aspirate (BMA) and the other side is local autograft combined with BMA. Therefore, all results per patient are the same results. All level results are the same unless specifically indicated, "per side".
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 29
units on a scale
  Baseline | 58.8 (26.2)
  6 Months: number analyzed (Participants) | 23
  6 Months | 79.2 (15.6)
  12 Months: number analyzed (Participants) | 16
  12 Months | 77.4 (17.0)
  24 Months: number analyzed (Participants) | 7
  24 Months | 72.9 (21.1)

6. Secondary Outcome: Number of Posterolateral Levels With Correlation of Fusion Ratings by X-ray and CT Scan
Description: Correlation of x-ray with computed tomography scan analysis at the 12 month follow-up time point.
Time Frame: 12 months
Measure: Count of Units; unit: Posterolateral Gutters
Units Other Than Participants: Posterolateral Gutters
Arm/Group | All Patients
Number analyzed (Participants) | 22
Number analyzed (Posterolateral Gutters) | 40
Posterolateral Gutters
  OsteoStrux (symptomatic): Agree | 37
  OsteoStrux (symptomatic): Disagree | 3
  Local Autograft (contralateral): Agree | 32
  Local Autograft (contralateral): Disagree | 8

7. Secondary Outcome: Medical Outcomes: Oswestry Disability Index (ODI), at All Available Time-points.
Description: The ODI is an index derived from the Oswestry Low Back Pain Questionnaire used by surgeons, clinicians and researchers to quantify disability for low back pain. The questionnaire is self-completed and covers 10 topics about pain intensity, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Scores are from 0-100 and a lower score represents a better score.
Time Frame: upto 24 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 29
units on a scale
  Baseline | 50.0 (17.3)
  6 Months: number analyzed (Participants) | 27
  6 Months | 39.3 (24.6)
  12 Months: number analyzed (Participants) | 23
  12 Months | 34.6 (22.7)
  24 Months: number analyzed (Participants) | 10
  24 Months | 33.7 (25.4)

8. Secondary Outcome: Medical Outcomes: Worst Leg Pain on the Visual Analog Scale (VAS) at All Available Time-points.
Description: The visual analogue scale (VAS) is a commonly used outcome measure for research studies. It is presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "0"/no pain at all" and "100/worst pain imaginable."
  The study in this scale is used for the worst leg pain. A lower score represents a better score.
Time Frame: upto 24 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Patients: All Patients
Arm/Group | All Patients
Number analyzed (Participants) | 24
units on a scale
  Baseline | 73.9 (21.6)
  6 Months | 30.5 (34.0)
  12 Months | 29.8 (34.3)
  24 Months | 24.4 (30.4)

9. Secondary Outcome: Medical Outcomes: Visual Analog Scale (VAS) Back Pain at All Available Time-points.
Description: The visual analogue scale (VAS) is a commonly used outcome measure for research studies. It is presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "0"/no pain at all" and "100/worst pain imaginable."
  The study in this scale is used for back pain. A lower score represents a better score.
Time Frame: upto 24 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 29
units on a scale
  Baseline | 70.2 (25.5)
  6 Months | 34.7 (30.9)
  12 Months | 32.3 (298)
  24 Months | 28.1 (18.5)

10. Secondary Outcome: Medical Outcomes: Maintenance of Lower Extremity Neurological Function at All Available Time-points.
Description: Posterolateral fusion study in which one spinal level is treated with both the study and control arm. The symptomatic posterolateral spinal side is OsteoStrux and the contralateral posterolateral spinal side is local autograft.
  NA (Not Applicable): Neurological function data was not able to be analyzed as there was a limitation of the method in the ability to distinguish between posterolateral sides in a neurological function assessment. Neurological function is indistinguishable between the right and left posterolateral sides of the lower extremities using the methods in the protocol. Therefore, this outcomes measure was not applicable.
Time Frame: upto 24 months
Population: NA (Not Applicable): Neurological function data was not able to be analyzed as there was a limitation of the method in the ability to distinguish between posterolateral sides in a neurological function assessment.
Groups:
- All Patients: Posterolateral fusion study in which one spinal level is treated with both the study and control arm. The symptomatic posterolateral spinal side is OsteoStrux and the contralateral posterolateral spinal side is local autograft.
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: Serious Adverse Events, Adverse Device Effects, Serious Adverse Device Effects and Subsequent surgical interventions.
Groups:
- All Patients: Posterolateral fusion study in which each patient undergoes posterolateral fusion. During the posterolateral fusion, each spinal level is treated with two grafts, the symptomatic posterolateral gutter is treated with study arm (OsteoStrux) and the contralateral posterolateral gutter is treated with the control arm (local autograft). Adverse events are unable to be distinguished per posterolateral gutter or spinal level and therefore results are submitted on a per patient basis.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 5/29
Other Adverse Events (participants affected / at risk) | 3/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=29)
bilateral hip replacement (Surgical and medical procedures) | 1 (1)
renal insufficiency (Endocrine disorders) | 1 (1)
hip infection after hip replacement (Infections and infestations) | 1 (1)
cage migration secondary to poor bone quality which required revision (Surgical and medical procedures) | 1 (1)
one episode of increased pain in low back and both legs which required hospitalization w/out surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
one episode of self-admittance to hospital for 8 days to detox from medication (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=29)
Small Durotomy/Dural Tear (Surgical and medical procedures) | 3 (3)

LIMITATIONS AND CAVEATS:
The following outcomes were unable to be analyzed due to the limitations of the protocol and analysis design and the inability to distinguish differences in posterolateral gutter analysis; neurological function and interbody fusion assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No